CLINICAL TRIAL: NCT03946267
Title: Infracyanine Green vs Brilliant Blue G in Inverted Flap Surgery for Medium to Large Macular Holes: A Swept Source OCT Analysis.
Brief Title: Infracyanine Green vs Brilliant Blue G in Macular Hole Inverted Flap Surgery: A Swept Source OCT Analysis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo (Other)
Responsible Party: Principal Investigator, Salvatore Cillino, Head of the Ophthalmology Section of the Department of Biomedicine, Neurosciences and Advanced Diagnostic, Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11/2016
Record Dates: First submitted 2019-05-09; First posted 2019-05-10 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Macular Holes
Keywords: Large macular hole; Inverted flap surgery; Infracyanine green; Brilliant blue G; Swept source OCT
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Intervention Model Description: Patients assigned to undergo inverted flap surgery with infracyanine green or with brilliant blue G using the sealed-envelope randomization technique. The interventional study model consists of a randomized controlled trial study design.
Who Masked: Participant, Outcomes Assessor
Masking Description: Authors involved in clinical data collection and measurement of outcome variables are not been directly involved in the patients' surgery and are masked to the randomization process
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IFCG = Infracyanine Green stained eyes (Experimental): After removal of core and posterior cortical vitreous and hyaloid stained with 0.2 ml triamcinolone acetonide 40 mg/mL, on the basis of the previous randomization the ILM is stained with 0.2 ml of low-concentration (0.5 mg/mL, 0.05%) IFCG injected over the macular area with the infusion line closed.
  Interventions: Device: Inverted inner limiting membrane flap technique for large full thickness macular holes
- BBG = Brilliant Peel stained eyes (Experimental): After removal of core and posterior cortical vitreous and hyaloid stained with 0.2 ml triamcinolone acetonide 40 mg/mL, on the basis of the previous randomization the ILM is stained with 0.2 mL BBG at a concentration of 0.25 mg/mL (0.025%) injected over the macular area with the infusion line closed.
  Interventions: Device: Inverted inner limiting membrane flap technique for large full thickness macular holes

INTERVENTIONS:
Device: Inverted inner limiting membrane flap technique for large full thickness macular holes — The ILM, stained with IFCG or BBG, is peeled off with ILM forceps, usually beginning near the inferotemporal vascular arcade, at least 2 disk diameters from the macular hole, in a circular manner. The peeling is extended up to the edges of the macular hole, the wide ILM flap obtained reduced by trimming with the vitreous cutter, and the annular remnant of ILM hinged to the hole's edge gently inverted upside down facing the RPE. Therefore, the hole is covered with usually more layers of inverted ILM. Attention is paid to avoid insertion and filling of the hole volume with ILM.

SUMMARY:
This study will compare by swept-source optical coherence tomography (SS-OCT) the retinal morphology after inverted internal limiting membrane (I-ILM) flap vitreoretinal surgery for medium-to-large macular holes using infracyanine green (IFCG) vs brilliant blue G (BBG) dyeing. It is a single-center prospective, randomized study. One group of patients will undergo I-ILM vitrectomy with IFCG staining, the other vitrectomy with BBG staining. Postoperative twelve-month corrected distance visual acuity, macular hole closure rate, and SS-OCT parameters will be compared and statistically analyzed. The aim of the study is to verify if these parameters can be negatively affected by toxicity related to the use of one of the two dyes.

DETAILED DESCRIPTION:
The purpose of this study is to compare by swept-source optical coherence tomography (SS-OCT) the retinal morphology after inverted internal limiting membrane flap (I-ILM) surgery for medium-to-large macular holes (FTMHs) using infracyanine green (IFCG) vs brilliant blue G (BBG). This prospective randomized study include 40 eyes with ≥ 400 µ idiopathic FTMH undergoing IFCG or BBG-stained I-ILM technique. Just before surgery, randomization is performed using the sealed-envelope technique, based on the patients' surgical chart number. The random allocation sequence is generated by the trial statistician pulling 41 standard-sized pieces of paper out of a hat. Twenty pieces of paper are marked with the Letter I, for IFCG, and 21 with the Letter B, for BBG. The trial statistician then sequentially puts each piece of paper into 41 sealed opaque envelopes. These envelopes are numbered 1 to 41 and given to the surgeons. Patients are numbered randomly from 1 to 41 based on a surgical chart number related to the baseline testing session and intervention period. Clinical data collection and measurement of outcome variables are performed by personnel masked to the randomization process and not been directly involved in the patients' surgery.

ELIGIBILITY:
Inclusion Criteria:

* Phakic or pseudophakic patients affected with medium to large idiopathic full thickness macular hole (FTMH), with a minimum preoperative diameter of 400 µ

Exclusion Criteria:

* Patients with chorioretinal diseases except FTMH, myopia > 5 D, history of glaucoma, previous trauma or ocular surgery other than cataract extraction, or conditions affecting visual acuity except cataract.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
Postoperative macular hole closure rate and morphology | twelve months
  Evaluated by swept-source OCT (Topcon DRI OCT Triton Series)
Postoperative mean corrected distance visual acuity | twelve months
  measured in logMAR notation using Early Treatment of Diabetic Retinopathy Study charts (CC-100XP LCD System for ETDRS Chart display)
Postoperative sizes of ellipsoid zone (EZ) and external limiting membrane (ELM) defects | twelve months
  Measured in micrometers by three-dimensional (3D) volumetric scan with swept-source OCT (Topcon DRI OCT Triton Series)
Thickness maps of the 1 mm central foveal thickness; second 3-mm grid including parafoveal macular area; second and the third 6-mm grid including parafoveal and perifoveal ganglion cells and inner plexiform layer; peripapillary nerve fiber layer. | twelve months
  Measured in micrometers by auto-segmentation software (Topcon Advanced Boundary Software - TABSTM)

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Cillino, MD, PhD, Principal Investigator — AOUP Paolo Giaccone, Palermo
Locations (1):
- Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Michalewska Z, Michalewski J, Adelman RA, Nawrocki J. Inverted internal limiting membrane flap technique for large macular holes. Ophthalmology. 2010 Oct;117(10):2018-25. doi: 10.1016/j.ophtha.2010.02.011. Epub 2010 Jun 11. PMID 20541263
- [Background] Haritoglou C, Tadayoni R, May CA, Gass CA, Freyer W, Priglinger SG, Kampik A. Short-term in vivo evaluation of novel vital dyes for intraocular surgery. Retina. 2006 Jul-Aug;26(6):673-8. doi: 10.1097/01.iae.0000236505.42892.54. PMID 16829811
- [Background] Schmid-Kubista KE, Lamar PD, Schenk A, Stolba U, Binder S. Comparison of macular function and visual fields after membrane blue or infracyanine green staining in vitreoretinal surgery. Graefes Arch Clin Exp Ophthalmol. 2010 Mar;248(3):381-8. doi: 10.1007/s00417-009-1213-4. Epub 2009 Oct 13. PMID 19823863
- [Background] Burk SE, Da Mata AP, Snyder ME, Rosa RH Jr, Foster RE. Indocyanine green-assisted peeling of the retinal internal limiting membrane. Ophthalmology. 2000 Nov;107(11):2010-4. doi: 10.1016/s0161-6420(00)00375-4. PMID 11054324
- [Background] Iriyama A, Uchida S, Yanagi Y, Tamaki Y, Inoue Y, Matsuura K, Kadonosono K, Araie M. Effects of indocyanine green on retinal ganglion cells. Invest Ophthalmol Vis Sci. 2004 Mar;45(3):943-7. doi: 10.1167/iovs.03-1026. PMID 14985315
- [Background] Baba T, Hagiwara A, Sato E, Arai M, Oshitari T, Yamamoto S. Comparison of vitrectomy with brilliant blue G or indocyanine green on retinal microstructure and function of eyes with macular hole. Ophthalmology. 2012 Dec;119(12):2609-15. doi: 10.1016/j.ophtha.2012.06.048. Epub 2012 Aug 24. PMID 22921387
- [Background] Park JH, Lee SM, Park SW, Lee JE, Byon IS. Comparative analysis of large macular hole surgery using an internal limiting membrane insertion versus inverted flap technique. Br J Ophthalmol. 2019 Feb;103(2):245-250. doi: 10.1136/bjophthalmol-2017-311770. Epub 2018 Apr 2. PMID 29610221